CLINICAL TRIAL: NCT00558285
Title: A Randomized, Double Blind, Placebo Controlled, Multicenter Study to Determine the Effect of QVA149 on Mean 24-hours Heart Rate in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Safety and Tolerability of QVA149 (Indacaterol/Glycopyrrolate) Compared to Placebo and to Indacaterol in Patients With Moderate to Severe Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149A2203
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Indacaterol; QVA149
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Glycopyrrolate; indacaterol-glycopyrronium combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- indacaterol/glycopyrrolate 600/100 μg (Experimental): Two capsules indacaterol/glycopyrrolate 300/50 μg delivered via a single dose dry powder inhaler in the morning for 14 days.
  The use of salbutamol/albuterol as rescue medication was permitted throughout the study.
  Interventions: Drug: indacaterol/glycopyrrolate
- indacaterol/glycopyrrolate 300/100 μg (Experimental): One capsule indacaterol/glycopyrrolate 300/100 μg and one placebo capsule delivered via a single dose dry powder inhaler in the morning for 14 days.
  The use of salbutamol/albuterol as rescue medication was permitted throughout the study.
  Interventions: Drug: indacaterol/glycopyrrolate; Drug: placebo
- indacaterol/glycopyrrolate 150/100 μg (Experimental): One capsule indacaterol/glycopyrrolate 150/50 μg and one capsule 50 μg glycopyrrolate delivered via a single dose dry powder inhaler in the morning for 14 days.
  The use of salbutamol/albuterol as rescue medication was permitted throughout the study.
  Interventions: Drug: indacaterol/glycopyrrolate; Drug: glycopyrrolate
- indacaterol 300 μg (Active Comparator): One capsule indacaterol 300 μg and one placebo capsule delivered via s single dose dry powder inhaler in the morning for 14 days.
  The use of salbutamol/albuterol as rescue medication was permitted throughout the study.
  Interventions: Drug: indacaterol; Drug: placebo
- placebo (Placebo Comparator): Two placebo capsules delivered via a single dose dry powder inhaler in the morning for 14 days.
  The use of salbutamol/albuterol as rescue medication was permitted throughout the study.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: indacaterol/glycopyrrolate — Inhalation capsule delivered via a single dose dry powder inhaler in the morning for 14 days.
  Other Names: QVA149
  Arms: indacaterol/glycopyrrolate 150/100 μg; indacaterol/glycopyrrolate 300/100 μg; indacaterol/glycopyrrolate 600/100 μg
Drug: indacaterol — Inhalation capsule delivered via a single dose dry powder inhaler in the morning for 14 days.
  Other Names: QAB149
  Arms: indacaterol 300 μg
Drug: glycopyrrolate — Inhalation capsule delivered via a single dose dry powder inhaler in the morning for 14 days.
  Arms: indacaterol/glycopyrrolate 150/100 μg
Drug: placebo — Inhalation capsule delivered via a single dose dry powder inhaler in the morning for 14 days.
  Arms: indacaterol 300 μg; indacaterol/glycopyrrolate 300/100 μg; placebo

SUMMARY:
An investigational inhalation product (QVA149) for the treatment of patients with Chronic Obstructive Pulmonary Disease (COPD) is being developed. This 14 day study will investigate the effect on heart rate and cardiovascular effects to ensure the product is safe.

ELIGIBILITY:
Inclusion Criteria:

* Consented male or female adults aged ≥40 years
* Moderate to severe stable Chronic Obstructive Pulmonary Disease (COPD) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines (2006)
* Patients who have smoking history of at least 10 pack years
* Patients with a post-bronchodilator Forced Expiratory Volume in one second (FEV1) ≥30% and <80% of the predicted normal and post-bronchodilator FEV1/Forced vital capacity (FVC) <0.70 at Visit 1 and Visit 3

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Patients requiring long term oxygen therapy (> 15 hours a day) on a daily basis for chronic hypoxemia, or who have been hospitalized or visited an emergency room for a COPD exacerbation in the 6 weeks prior to screening (Visit 1) or during the screening period
* Patients who had a respiratory tract infection within 6 weeks of Visit 1 or at screening
* Concomitant pulmonary disease, pulmonary tuberculosis (TB) (unless chest x-ray confirms no longer active) or clinically significant bronchiectasis
* Any history of asthma
* Patients who have clinically relevant lab abnormalities / conditions such as (but not limited to) long term prednisone therapy, unstable ischemic heart disease, left ventricular failure, history of myocardial infarction, arrhythmia (excluding stable atrial fibrillation [AF]), uncontrolled hypertension, narrow-angle glaucoma, symptomatic prostatic hyperplasia or bladder-neck obstruction or moderate to severe renal impairment, uncontrolled hypo- and hyperthyroidism, hypokalemia, hyperadrenergic state or any condition which might compromise patient safety or compliance, interfere with evaluation, or preclude completion of the study
* Patients with a history of cardiac failure, life threatening arrhythmias (screening Holter) and acute ischemic changes (screening ECG)
* Patients with a history of long QT syndrome or whose QTc (Fridericia method) interval measured at screening (Visit 1) is prolonged (>450 ms for males or >470 for females)
* History of malignancy of any organ system, treated or untreated within the past 5 years
* Uncontrolled Type I / Type II Diabetes or blood glucose outside the normal range or Hemoglobin A1C (HbA1c) >8.0% of total hemoglobin measured at Visit 1

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Novartis Pharmaceuticals
Locations (40):
- Australia (5):
  - Novartis Investigator Site, Adelaide
  - Novartis Investigator Site, Clayton
  - Novartis Investigator Site, Daw Park
  - Novartis Investigator site, Heidelberg
  - Novartis Investigator Site, Nedlands
- Belgium (5):
  - Novartis Investigator Site, Brussels
  - Novartis Investigator Site, Jambes
  - Novartis Investigator Site, Jette
  - Novartis Investigator site, Liège
  - Novartis Investigator Site, Ostend
- Canada (6):
  - Novartis Investigator Site, Mississauga
  - Novartis Investigator Site, Newmarket
  - Novartis Investigator Site, Ottawa
  - Novartis Investigator Site, Pointe-Claire
  - Novartis Investigator Site, Québec
  - Novartis Investigator Site, Sainte-Foy
- France (7):
  - Novartis Investigator Site, Ambroise
  - Novartis Investigator Site, Lille
  - Novartis Investigator Site, Marseille
  - Novartis investigator site, Martigues
  - Novartis Investigator Site, Nantes
  - Novartis Investigator site, Nice
  - Novartis Investigator Site, Perpignan
- Germany (6):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Dortmund
  - Novartis Investigator Site, Erfurt
  - Novartis Investigator Site, Hanover
  - Novartis Investigator Site, Mainz
  - Novartis Investigator Site, Marburg
- Italy (3):
  - Novartis Investigator Site, Florence
  - Novartis Investigator site, Modena
  - Novartis Investigator Site, Trieste
- Spain (6):
  - Novartis Investigator Site, Badalona
  - Novartis Investigator Site, Barakaldo
  - Novartis Investigator Site, Cáceres
  - Novartis Investigator Site, Centelles
  - Novartis Investigator Site, Mataró
  - Novartis Investigator Site, Valencia
- Turkey (Türkiye) (2):
  - Novartis Investigator Site, Istanbul
  - Novartis Investigator Site, Izmir

RESULTS

PARTICIPANT FLOW:
Groups:
- Indacaterol/Glycopyrrolate 600 μg/100 μg: Two capsules indacaterol/glycopyrrolate 300 μg/50 μg delivered via a single dose dry powder inhaler in the morning for 14 days.
  The use of salbutamol/albuterol as rescue medication was permitted throughout the study.
- Indacaterol/Glycopyrrolate 300 μg/100 μg: One capsule indacaterol/glycopyrrolate 300 μg/100 μg and one placebo capsule delivered via a single dose dry powder inhaler in the morning for 14 days.
  The use of salbutamol/albuterol as rescue medication was permitted throughout the study.
- Indacaterol/Glycopyrrolate 150 μg/100 μg: One capsule indacaterol/glycopyrrolate 150 μg/50 μg and one capsule 50μg glycopyrrolate delivered via a single dose dry powder inhaler in the morning for 14 days.
  The use of salbutamol/albuterol as rescue medication was permitted throughout the study.
Period: Overall Study
Arm/Group | Indacaterol/Glycopyrrolate 600 μg/100 μg | Indacaterol/Glycopyrrolate 300 μg/100 μg | Indacaterol/Glycopyrrolate 150 μg/100 μg | Indacaterol 300 μg | Placebo
Started | 50 | 51 | 51 | 52 | 53
Safety: Received Study Drug | 49 | 51 | 51 | 51 | 53
Completed | 44 | 48 | 46 | 48 | 49
Not Completed | 6 | 3 | 5 | 4 | 4
Not completed — Adverse Event | 1 | 1 | 4 | 1 | 2
Not completed — Abnormal test procedure result(s) | 1 | 0 | 0 | 0 | 0
Not completed — Subject withdrew consent | 2 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Administrative problems | 0 | 0 | 0 | 1 | 1
Not completed — Protocol deviation | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol/Glycopyrrolate 600/100 μg | Indacaterol/Glycopyrrolate 300/100 μg | Indacaterol/Glycopyrrolate 150/100 μg | Indacaterol 300 μg | Placebo | Total
Number analyzed (Participants) | 49 | 51 | 51 | 51 | 53 | 255
Age Continuous [Mean (Standard Deviation); unit: years] — Overall Number of Baseline Participants is based on the Safety Population
  years | 65.7 (9.34) | 63.7 (8.94) | 60.9 (8.58) | 64.5 (9.75) | 64.3 (8.95) | 63.8 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 15 | 10 | 14 | 60
  Male | 38 | 41 | 36 | 41 | 39 | 195

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean 24 Hour Heart Rate at Day 14
Description: Heart rate was assessed by Holter monitoring and was measured over a 24 hour period at day 14. Heart rate was defined as the average value over the 24 hour monitoring period. The baseline measurement was the average heart rate taken from the 24 hour Holter monitoring period performed at screening or the last 24-hour period before taking the first dose of study drug. Least square means are based on the analysis of covariance: 24 hours mean heart rate = center + treatment + baseline value + Forced Expiratory Volume in one second (FEV1) before inhalation of salbutamol/albuterol + FEV1 30 min post salbutamol/albuterol + error.
Time Frame: Baseline, Day 14
Population: Safety Population includes all patients who received at least one dose of study drug. Participants with less than 18 hours quality recording time data were excluded from this analysis.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Indacaterol/Glycopyrrolate 600/100 μg | Indacaterol/Glycopyrrolate 300/100 μg | Indacaterol/Glycopyrrolate 150/100 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 39 | 45 | 40 | 42 | 45
beats per minute | -0.113 (0.9967) | 0.787 (0.8975) | -0.230 (0.9567) | 0.240 (0.9373) | 0.170 (0.8760)

2. Secondary Outcome: Change From Baseline in Mean 24 Hour Heart Rate at Day 1
Description: Heart rate was assessed by Holter monitoring and was measured over a 24 hour period at day 1. Heart rate was defined as the average value over the 24 hour monitoring period. The baseline measurement was the average heart rate taken from the 24 hour Holter monitoring period performed at screening or the last 24-hour period before taking the first dose of study drug. Least squares means are based on the analysis of covariance: 24 hours mean heart rate = center + treatment + baseline value + Forced Expiratory Volume in one second (FEV1) before inhalation of salbutamol/albuterol + FEV1 30 min after inhalation of salbutamol/albuterol + error.
Time Frame: Baseline, Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Indacaterol/Glycopyrrolate 600/100 μg | Indacaterol/Glycopyrrolate 300/100 μg | Indacaterol/Glycopyrrolate 150/100 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 45 | 46 | 47 | 48 | 47
beats per minute | -2.877 (0.8790) | -2.770 (0.8244) | -0.547 (0.8208) | -1.849 (0.8211) | -0.329 (0.8181)

3. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Day 1 and Day 14
Description: Spirometry testing was performed in accordance with American Thoracic Society standards. Trough FEV1 was defined as the mean of two measurements at 23 hours 15 minutes and 23 hour 45 minutes post dosing. Baseline is defined as the mean of the two values taken at 45 minutes and 15 minutes prior to dosing at day 1. Least square means are based on the analysis of covariance: response variable=center + treatment + baseline value + Forced Expiratory Volume in one second (FEV1) before inhalation of salbutamol/albuterol + FEV1 30 minutes post inhalation of salbutamol/albuterol.
Time Frame: Day 1, Day 14
Population: Intent-to-treat Population includes all randomized patients. Any spirometric data collected less than six hours after rescue medication use was regarded as missing.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol/Glycopyrrolate 600/100 μg | Indacaterol/Glycopyrrolate 300/100 μg | Indacaterol/Glycopyrrolate 150/100 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 50 | 51 | 51 | 52 | 53
Liters
  Day 1 | 1.59 (0.024) | 1.51 (0.023) | 1.50 (0.022) | 1.44 (0.023) | 1.27 (0.022)
  Day 14 | 1.61 (0.027) | 1.52 (0.025) | 1.50 (0.026) | 1.46 (0.025) | 1.31 (0.024)

4. Secondary Outcome: Trough Forced Vital Capacity (FVC) at Day 1 and Day 14
Description: Spirometry testing was performed in accordance with American Thoracic Society standards. Trough FVC was defined as the mean of two measurements at 23 hours 15 minutes and the 23 hours 45 minutes post dosing. Baseline was defined as the mean of the two values taken at 45 minutes and 15 minutes prior to dosing at day 1. Analysis of covariance: FVC parameter = center + treatment + baseline FVC + FEV1 before inhalation of salbutamol/albuterol + FEV1 30 min after inhalation of salbutamol/albuterol + error.
Time Frame: Day 1 and Day 14
Population: Participants from the Intent-to-treat Population (all randomized patients) with data available at the given time-point. Any spirometric data collected less than six hours after rescue medication use was regarded as missing.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol/Glycopyrrolate 600/100 μg | Indacaterol/Glycopyrrolate 300/100 μg | Indacaterol/Glycopyrrolate 150/100 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 48 | 48 | 51 | 49 | 52
Liters
  Day 1 | 3.151 (0.0437) | 3.029 (0.0421) | 3.000 (0.0403) | 2.924 (0.0419) | 2.634 (0.0402)
  Day 14 (n=42, 45, 44, 48, 47) | 3.134 (0.0469) | 3.042 (0.0446) | 2.952 (0.0455) | 2.901 (0.0442) | 2.726 (0.0424)

5. Secondary Outcome: Change From Baseline in QTc (Fridericia's Formula) at Day 1
Description: The change from baseline in QTc at 30 minutes, 4 hours and 23 hours 45 minutes post dose on day 1. QT calculated (QTc) was calculated from the QT interval and RR (in seconds) using Fridericia's formula: QTc = QT / 3√ RR. Least square means are based on the analysis of covariance: response variable = center + treatment + baseline value + FEV1 before inhalation of salbutamol/albuterol + FEV1 30 min post inhalation of salbutamol/albuterol.
Time Frame: Baseline, Day 1
Population: Safety Population includes all patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Indacaterol/Glycopyrrolate 600/100 μg | Indacaterol/Glycopyrrolate 300/100 μg | Indacaterol/Glycopyrrolate 150/100 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 49 | 51 | 51 | 51 | 53
milliseconds
  30 minutes | 1.6 (1.58) | 1.2 (1.48) | 1.4 (1.50) | 3.1 (1.47) | -1.6 (1.44)
  4 hours | 2.8 (1.67) | 0.5 (1.56) | 2.4 (1.58) | 1.1 (1.60) | -2.3 (1.52)
  23 hours 45 minutes | 2.7 (1.77) | -1.7 (1.66) | -0.1 (1.67) | -2.1 (1.71) | -2.3 (1.62)

6. Secondary Outcome: Change From Baseline in QTc (Fridericia's Formula) at Day 7
Description: The change from baseline in QTc at 30 minutes and 2 hours post dose on day 7. QT calculated (QTc) was calculated from the QT interval and RR (in seconds) using Fridericia's formula: QTc = QT / 3√ RR. Least square means are based on the analysis of covariance: response variable = center + treatment + baseline value + FEV1 before inhalation of salbutamol/albuterol + FEV1 30 min post inhalation of salbutamol/albuterol.
Time Frame: Baseline, Day 7
Population: Safety Population includes all patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Indacaterol/Glycopyrrolate 600/100 μg | Indacaterol/Glycopyrrolate 300/100 μg | Indacaterol/Glycopyrrolate 150/100 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 49 | 51 | 51 | 51 | 53
milliseconds
  30 minutes | 4.1 (1.91) | -0.9 (1.74) | 0.5 (1.78) | -1.3 (1.79) | -2.2 (1.70)
  2 hours | 2.6 (2.17) | -1.2 (1.98) | 1.6 (2.02) | -1.6 (2.00) | -2.8 (1.94)

7. Secondary Outcome: Change From Baseline in QTc (Fridericia's Formula) at Day 14
Description: The change from baseline in QTc at 30 minutes, 4 hours and 23 hours 45 minutes post dose on day 14. QT calculated (QTc) was calculated from the QT interval and RR (in seconds) using Fridericia's formula: QTc = QT / 3√ RR. Least square means are based on the analysis of covariance: response variable = center + treatment + baseline value + FEV1 before inhalation of salbutamol/albuterol + FEV1 30 minutes post inhalation of salbutamol/albuterol.
Time Frame: Baseline, Day 14
Population: Safety Population includes all patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Indacaterol/Glycopyrrolate 600/100 μg | Indacaterol/Glycopyrrolate 300/100 μg | Indacaterol/Glycopyrrolate 150/100 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 49 | 51 | 51 | 51 | 53
milliseconds
  30 minutes | 2.4 (1.79) | -0.6 (1.64) | 1.6 (1.70) | -1.2 (1.69) | 0.2 (1.62)
  4 hours | 2.8 (1.90) | -0.1 (1.76) | 3.1 (1.85) | -2.6 (1.81) | -0.1 (1.73)
  23 hours 45 minutes | 0.5 (1.94) | -2.9 (1.81) | 0.4 (1.95) | -3.6 (1.88) | -1.6 (1.77)

ADVERSE EVENTS:
Groups:
- Placebo: Two placebo capsules delivered via a single dose dry powder inhaler in the morning for 14 days.
  The use of salbutamol /albuterol as rescue medication was permitted throughout the study.
Arm/Group | Indacaterol/Glycopyrrolate 600/100 μg | Indacaterol/Glycopyrrolate 300/100 μg | Indacaterol/Glycopyrrolate 150/100 μg | Indacaterol 300 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/49 | 0/51 | 2/51 | 0/51 | 1/53
Other Adverse Events (participants affected / at risk) | 5/49 | 6/51 | 10/51 | 7/51 | 4/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol/Glycopyrrolate 600/100 μg (N=49) | Indacaterol/Glycopyrrolate 300/100 μg (N=51) | Indacaterol/Glycopyrrolate 150/100 μg (N=51) | Indacaterol 300 μg (N=51) | Placebo (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol/Glycopyrrolate 600/100 μg (N=49) | Indacaterol/Glycopyrrolate 300/100 μg (N=51) | Indacaterol/Glycopyrrolate 150/100 μg (N=51) | Indacaterol 300 μg (N=51) | Placebo (N=53)
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 3 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 2 | 3 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 2 | 1
Hypertension (Vascular disorders) | 0 | 3 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.